CLINICAL TRIAL: NCT03877016
Title: Prospective, Multicentric, Randomized on Two Arms, Controlled, by Cross-over, Pilot Study, in Order to Evaluate Disconfort Among Outpatients Using actiTENS for Neuropathic Pain vs TENS ECO 2.
Brief Title: Pilot Study in Order to Evaluate Disconfort Among Outpatients Using actiTENS for Neuropathic Pain vs TENS ECO 2.
Acronym: QolTENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PI2018_843_0028
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Neuropathic Pain
Keywords: neuropathic pain; electrical nerve stimulation therapy; patient report outcomes; non-pharmalogical treatment
MeSH Terms: conditions — Neuralgia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS Eco2 (Active Comparator): TENS Eco2 is the classical device in patients with chronic neuropathic pain
  Interventions: Procedure: TENS
- actiTENS (Experimental): ActiTENS is a new TENS device, that seems less cotraining.
  Interventions: Procedure: TENS

INTERVENTIONS:
Procedure: TENS — TENS Eco2 or actiTENS, both admitted and reimbursed in FRANCE according to regulation

SUMMARY:
Non-pharmacological treatments for pain relief are more and more used in clinical care although any scientific validation. Among the non-pharmacological treatments of neuropathic pain relief, TENS (Electrical Nerve Stimulation Therapy) is the major treatment with the best benefit. Unfortunately, the use of TENS by patients appears very difficult. Because of this inconvenience, more than 40% of TENS users interrupt the treatment despite treatment benefit. A new TENS device: actiTENS that seems to be less constraining than TENS is now available in France. ActiTENS efficacy and safety compared to TENS need to be investigated.

The main objective is to evaluate and to compare the use of actiTENS, with TENS Eco 2, the classical device in patients with chronic neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Patient covered by national health insurance
* Patient able to express consent
* Patient with neuropathic pain with DN4 (Douleur Neuropathique 4 Questions) > or = 4/10.
* Actual or potential neurologic lesion
* Patient still using a TENS device

Exclusion Criteria:

* Planned surgery in the next two months
* Modification of the reatment in the next two motnhs
* Other study ongoing for the patient
* Medical contraindication for TENS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Disconfort of using TENS (Electrical Nerve Stimulation Therapy) Eco2 versus actiTENS | day7 after patient inclusion
  Discomfort evaluation will be determined by using VAS (Visual Analogue Scale)
Disconfort of using TENS (Electrical Nerve Stimulation Therapy) Eco2 versus actiTENS | day 35 after patient inclusion
  Discomfort evaluation will be determined by using VAS (Visual Analogue Scale)

SECONDARY OUTCOMES:
length of TENS daily use | day7 after patient inclusion
  Length of TENS daily use
length of TENS daily use | day 35 after patient inclusion
  Length of TENS daily use

CONTACTS AND LOCATIONS:
Overall Officials: Eric SERRA, MD, Principal Investigator — CHU Amiens
Locations (5):
- France (5):
  - CHU Amiens Picardie, Amiens
  - CHD La Roche Sur Yon, La Roche-sur-Yon
  - CHU de Nantes, Nantes
  - APHP - Hopital Saint Antoine, Paris
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No